CLINICAL TRIAL: NCT04300959
Title: Anlotinib Hydrochloride in Combination With PD1 With Gemcitabine Plus(+)Cisplatin Compared With Gemcitabine +Cisplatin as First-line Chemotherapy for Unresectable or Metastatic Biliary Tract Cancer: A Randomized, Controlled, Multicenter Phase II Clinical Trial
Brief Title: Anlotinib in Combination With PD1 With Gemcitabine Plus(+)Cisplatin for Unresectable or Metastatic Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTNZJ-004
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — anlotinib; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Anlotinib in combination with Sintilimab with Gemcitabine plus(+)Cisplatin
  Interventions: Drug: Anlotinib Hydrochloride in Combination With PD1 With Gemcitabine Plus(+)Cisplatin
- Control group (Active Comparator): Standard platinum-based chemotherapy
  Interventions: Drug: Gemcitabine Plus(+)Cisplatin

INTERVENTIONS:
Drug: Anlotinib Hydrochloride in Combination With PD1 With Gemcitabine Plus(+)Cisplatin — Gemcitabine:1000mg/m2, days 1 and 8; Cisplatin: 25mg/m2, days 1 and 8； Anlotinib : 10mg po qd, days 1-14; Sintilimab: 200mg IV, day 1；
  1 cycle = 3 weeks.
  Other Names: AL3818; IBI308
  Arms: Experimental group
Drug: Gemcitabine Plus(+)Cisplatin — Gemcitabine:1g/m2, days 1 and 8; Cisplatin: 25mg/m2, days 1 and 8；
  1 cycle = 3 weeks.
  Arms: Control group

SUMMARY:
To evaluate the efficacy and safety of Anlotinib Hydrochloride in Combination With PD1 With Gemcitabine Plus(+)Cisplatin Compared With Gemcitabine +Cisplatin as First-line Chemotherapy for Unresectable or Metastatic Biliary Tract Cancer

DETAILED DESCRIPTION:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and c-Kit kinase.It is a randomized, controlled, multicenter phase II clinical trial conducted in China, and plan to recruit 80 patients who were primarily diagnosed with unresectable or metastatic biliary tract cancer who have not received previous systemic treatment.To evaluate the efficacy and safety of Anlotinib Hydrochloride in Combination With PD1 With Gemcitabine Plus(+)Cisplatin Compared With Gemcitabine +Cisplatin as First-line Chemotherapy for Unresectable or Metastatic Biliary Tract Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are voluntary and sign an informed consent document.
2. Age between 18-70 years (including 18 and 70), no gender preference.
3. Expected survival ≥ 12 weeks
4. ECOG performance status 0 or 1 within 7 days prior to the first dose.
5. In women of child-bearing age, pregnancy test should be negative within 28 days prior to registration, and effective contraception during the treatment period should be adopted within 60 days after the last dose. In this trial, women of child-bearing age are defined as sexually mature women with: 1) no history of hysterectomy or bilateral ovariectomy; 2) natural menopause < continuous 24 months (amenorrhea after cancer treatment does not preclude fertility) (i.e., having menstruation at any time within preceding continuous 24 months); female spouses of male subjects who are of child-bearing age should also follow the above contraceptive requirements.
6. Adequate organ function.

   Blood test (no blood transfusion, no usage of G-CSF and no medication for correction within 14 days prior to screening):
   1. neutrophil count ≥ 1.5×109/L
   2. platelets ≥ 75×109/L
   3. hemoglobin ≥ 90g/L

      Biochemical test (no albumin transfusion within 14 days prior to screening):
   4. serum creatinine ≤ 1.5× upper limit normal (ULN), or creatinine clearance > 50 mL/min;
   5. total bilirubin ≤ 1.5×ULN (total bilirubin ≤ 3× ULN in patients with Gilbert syndrome);
   6. AST and ALT ≤ 2.5× ULN; for patients with hepatic metastases, AST and ALT ≤ 5× ULN;
   7. INR ≤ 2.3 or prothrombin time (PT) exceeding normal control range ≤ 6 seconds;
   8. urine protein < 2+ (if urine protein ≥ 2+, 24-hour urine protein quantitation could be considered, and if 24-hour urine protein quantitation < 1.0g, the patient can be included).

      Cardiac function:
   9. NYHA < grade 3;
   10. LCEF ≥ 50%;
7. In patients with active HBV infection: HBV-DNA should < 500 IU/mL (if measured by copy/ml, HBV-DNA should <2500 copy/mL); patients should be willing to receive antiviral therapy during the treatment period. Patients with positive HCV-DNA should receive antiviral therapy according to local guidelines with liver function ≤ CTCAE grade 1.
8. Patients should have adequate nutritional condition, i.e., BMI≥ 18 kg/m2, weight ≥ 40 kg, and albumin ≥ 3.0 g/dL.
9. Histologically and/or cytologically-confirmed diagnosis of local advanced or metastatic cholangiocarcinoma (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma and gallbladder carcinoma), which is incurable and unresectable.
10. Having at least one site of measurable lesion (RECIST Version 1.1). Target lesion of tumor progression within previous radiation filed or locally-treated area could be considered as measurable.

Exclusion Criteria:

Patients who meet any of the following conditions will be excluded from the trial:

1. Patients who previously received systemic treatment for advanced unresectable or metastatic cholangiocarcinoma will be excluded. Neoadjuvant or adjuvant therapy is acceptable if treatment is completed at least 6 months prior to randomization and shows no progression.
2. Patients suffering from other active malignancies within 5 years or coexisting with cholangiocarcinoma, except adequately treated localized neoplasms including, but not limited to: basal cell or squamous cell skin cancer, superficial bladder cancer, in situ prostate cancer, in situ cervical cancer, and in situ breast cancer.
3. Patients who are preparing for or have previously undergone organ or allogenic bone marrow transplantation.
4. Patients with symptomatic moderate or severe ascites requiring paracentesis and drainage (except patients with imaging showing mild ascites but no clinical symptoms); or patients with uncontrolled or moderate and severe pleural or pericardial effusion.
5. Patients who have a history of gastrointestinal hemorrhage within preceding 6 months or gastrointestinal hemorrhagic tendency, e.g., esophagogastric varices with a risk of hemorrhage, active peptic ulcer, fecal occult blood being continuously positive (if fecal occult blood is positive at baseline, reexamination can be considered; if reexamination is still positive, esophagogastroduodenoscopy (EGD) should be considered; if EGD indicates esophagogastric varices with a risk of hemorrhage, then the patient will be excluded).
6. Patients with hereditary or acquired bleeding tendency (e.g., coagulation dysfunction) or thrombophilia, e.g., hemophilia patients; or patients who are currently receiving or recently received (within preceding 10 days) full-dose anticoagulant or thrombolytic agents orally or by injection for therapeutic purposes (prophylactic usage of low-dose aspirin or low molecular heparin is acceptable).
7. Patients who are receiving or recently received (within preceding 10days) aspirin (>325 mg/d (maximum antiplatelet dose)) or dipyridamole, ticlopidine, clopidogrel and cilostazol.
8. Patients who have a history of thrombosis or embolism within preceding 6 months, including cerebrovascular events (transient ischemic attack, cerebral hemorrhage and cerebral infraction) and pulmonary embolism.
9. Patients with uncontrolled heart disease or relevant symptoms, e.g., (1) heart failure with NYHA > 2 (Appendix 5) or UCG showing LVEF <50%; (2) unstable angina; (3) a history of myocardial infraction within preceding 1 year; (4) supraventricular or ventricular arrhythmia with clinical significance indicating treatment or intervention; (5) QTc > 450ms (male); QTc > 470ms(female) (QTc is calculated by Fridericia law; if QTc is abnormal, it can be continuously measured 3 times with an interval of 2 minutes, taking the average).
10. Patients with hypertension uncontrolled by drug or treatment (SBP≥140 mmHg or DBP≥90 mmHg) (based on≥2 measurements and taking average); or patients with a history of hypertensive emergency or hypertensive encephalopathy.
11. Patients who have severe vascular diseases (e.g., aortic aneurysm requiring surgical repair or with recent peripheral arterial thrombosis) within preceding 6 months.
12. Patients with severe, unhealed or open wounds, and active ulcers or untreated fractures.
13. Patients who received major operation (except diagnosis) within preceding 4 weeks, or who are expected to receive major operation during the trial period.
14. Patients who are unable to swallow tablets, or with malabsorption syndrome or any condition that may affect gastrointestinal absorption.
15. Patients with aeroperitoneum that cannot be explained by puncture or recent surgery.
16. Patients with brain metastases before or at present
17. Patients suffering from uncontrolled systemic diseases including, but not limited to: diabetes, hypertension, pulmonary fibrosis, acute pulmonary disease, interstitial lung disease, cirrhosis, angina and severe arrhythmia.
18. Patients suffering from interstitial pneumonia or ILD, or with a history of interstitial pneumonia or ILD requiring hormone therapy, or with other pulmonary fibrosis，organic pneumonia(e.g., obliterative bronchiolitis), pneumoconiosis, drug-induced pneumonia and idiopathic pneumonia that may interfere with the diagnosis and management of immune-related pulmonary toxicity; or patients with CT image indicating active pneumonia or severely impaired pulmonary function during screening. Radiation pneumonia is acceptable in the radiation field. Patients with active tuberculosis will be excluded.
19. Patients suffering from active autoimmune disease or with a history of autoimmune disease that may recur (including, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism and hypothyroidism [patients controlled only by hormone replacement therapy are acceptable]) will be excluded; patients with dermatosis requiring no systemic treatment, including vitiligo, psoriasis and alopecia, are acceptable; patients win T1DM controlled by insulin therapy, or patients with completely-relieved childhood asthma requiring no intervention in adulthood are acceptable; patients with asthma requiring bronchodilator intervention will be excluded.
20. Patients who received immunosuppressive drug or systemic hormone therapy to achieve immunosuppression (prednisone>10mg/d or hormones of equivalent effects) within preceding 14 days.
21. Patients who received strong CYP3A4/CYP2C19 inducer including rifampin (and its analogs) and hypericum perforatum or strong CYP3A4/CYP2C19 inhibitor within preceding 14 days.
22. Patients who have a history of severe allergies to any monoclonal antibody or anti-angiogenic targeted drugs.
23. Patients who had severe infection within preceding 4 weeks including, but not limited to: infection, bacteremia and complications of severe pneumonia resulting in hospitalization; or patients who received therapeutic antibiotics orally or intravenously within preceding 2 weeks (prophylactic usage of antibiotics [e.g., prevention of urinary tract infection or exacerbation of COPD] is acceptable).
24. Patients with innate or acquired immunodeficiency (e.g., patients infected with HIV)
25. Patients who previously received anti-PD-1 therapy or other immunotherapies targeting PD-1/PD-L1, or tyrosine kinase inhibitor therapy.
26. Palliative radiotherapy for non-target lesions to control symptoms is acceptable, but should be completed at least 2 weeks prior with adverse events not recovering to ≤CTCAE grade 1
27. Patients who received attenuated live vaccine within preceding 28 day, or who are expected to receive the vaccine during sintilimab treatment or within 60 days after the last dose of sintilimab.
28. Patients who received anti-tumor cytotoxic chemotherapy, biotherapy (e.g., monoclonal antibody), immunotherapy (e.g., IL-2 or interferon) or other investigational drugs within 4 weeks prior to registration.
29. Patients with other factors that may affect the outcomes or lead to withdrawal (judged by the researcher), including alcohol abuse, drug abuse, other serious disease (including mental illness) requiring combined treatment, significantly abnormal laboratory test index, and family or society factors that may affect patient safety.
30. Patients who previously received antitumor therapy and prior toxicity has not recovered to CTCAE grade 0-1, aside from the following conditions:

    1. alopecia;
    2. hyperpigmentation;
    3. peripheral neurotoxicity recovered to < CTCAE grade 2;
    4. long-term toxicity caused by radiotherapy cannot recover (judged by the researcher).
31. Patients who have active tuberculosis(TB) and are receiving anti-TB therapy, or who received anti-TB therapy within 1 year prior to screening.
32. Patients who are pregnant or lactating. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
12 months OS rate | 360 days
  The definition of 12-months OS rate is the percentage of patients who had NOT has an event before or at 12 months

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 24 months after enrollment or study close
  OS is calculated from diagnosis to death or last follow-up time
Progress free survival (PFS) | up to 24 months after enrollment or study close
  PFS is defined as the time from the date of treatment to the first date of disease progression or death from any cause
Objective response rate(ORR) | up to 24 months after enrollment or study close
  Number of participants with partial response or complete response treating by anloitnib according to RESIST criteria v1.1.
Incidence of Treatment-Emergent 3/4 Adverse Events | up to 24 months after enrollment or study close
  Number and percentage of participants with Adverse Events (any Grade and Grade 3/4).

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Zhou S, Xu X, Zheng Q, Zhang F, Luo C, Li D, Sun X, Han Z, Wu W, Yan J, Shao Y, Zhang Y, Wu B, Wei Q, Wang X, Zhou Y, Sun W, Xu Q, Ying J. Sintilimab and anlotinib with gemcitabine plus cisplatin in advanced biliary tract cancer: SAGC a randomized phase 2 trial. Nat Commun. 2025 Jul 1;16(1):5559. doi: 10.1038/s41467-025-60119-3. PMID 40593475